CLINICAL TRIAL: NCT01094535
Title: MRCP With Secretin Stimulation for the Evaluation of Pancreatic Endocrine and Exocrine Function Following Surgical Resection for Pancreatic Adenocarcinoma
Brief Title: Secretin-enhanced Magnetic Resonance Cholangiopancreatography (S-MRCP) and Pancreatic Function Following Surgery
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Poor enrollment
Sponsor: Columbia University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: AAAC0218
Record Dates: First submitted 2010-03-25; First posted 2010-03-29 (Estimated); Last update posted 2015-04-06 (Estimated); Status verified 2015-04

CONDITIONS: Pancreatic Cancer
Keywords: Pancreatic adenocarcinoma; Synthetic human secretin; Secretin-enhanced MRCP; Pancreatic insufficiency; Endoscopic Pancreatic Function Test (ePFT); Endocrine pancreatic function test; Exocrine pancreatic function test
MeSH Terms: conditions — Pancreatic Neoplasms; Exocrine Pancreatic Insufficiency | interventions — Secretin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Secretin (Experimental): One-arm (open label): Synthetic Human Secretin. Patients will undergo four Secretin-enhanced magnetic resonance cholangiopancreatography (S-MRCP) evaluations.
  Interventions: Drug: Synthetic Human Secretin

INTERVENTIONS:
Drug: Synthetic Human Secretin — S-MRCP has recently emerged as a widely-accepted noninvasive technique to assess morphological changes in the pancreatic ducts, as well as functional secretory capacity of the gland. Twelve patients will each undergo four Secretin-enhanced magnetic resonance cholangiopancreatography (S-MRCP) evaluations, at a dose of 0.2 ucg/kg per exam, each S-MRCP will require 16-32 ucg of secretin (12 vials). Secretin, provided by the Repligen Corporation, will be administered by IV bolus injection over 30 seconds followed by a 30 second saline flush. The maximum dose of secretin will be 18.5 ucg.
  Other Names: RG1068

SUMMARY:
The aim of this study will be to determine whether secretin-enhanced MRCP (S-MRCP) as well as traditional magnetic resonance imaging (MRI) of the pancreas will allow the investigators to quantify the pancreas' ability to secrete hormones as well as digestive enzymes, both before and after surgery. The investigators hypothesize that S-MRCP will provide a novel non-invasive measure of pancreatic function.

DETAILED DESCRIPTION:
Surgical resection offers the only hope of cure for pancreatic adenocarcinoma. While perioperative mortality rates have declined in recent years, pancreatectomy is still associated with significant postoperative malnutrition, maldigestion, and glucose intolerance, mostly as a result of pancreatic insufficiency. Quantifying residual pancreatic function remains a challenge, but is essential in improving the survival and quality of life of pancreatic cancer patients. Secretin-enhanced magnetic resonance cholangiopancreatography (S-MRCP)has recently emerged as a widely-accepted noninvasive technique to assess morphological changes in the pancreatic ducts, as well as functional secretory capacity of the gland. The aim of our study is to evaluate S-MRCP as a means to assess pancreatic reserve in patients who will undergoing surgical resection for pancreatic carcinoma. As an adjunct to S-MRCP, we will also evaluate the concomitant use of dynamic MRI with contrast enhancement. This will be a prospective study of twelve patients who will undergo S-MRCP/MRI within 30 days of surgery and then at 3, 6, and 12 months post-operatively. Quantitative analysis of S-MRCP will include pancreatic duct diameter and volume before and after secretin administration. MRI will be analyzed for mean T1 signal intensity, total parenchymal volume, and gadolinium enhancement. These radiological parameters will be compared to clinical parameters of exocrine function(subjective reporting of steatorrhea and abdominal pain as well as levels of fecal elastase1 and fat soluble vitamins in stool samples) as well as endocrine function (fasting blood glucose, hemoglobin A1c, amylin, glucagon, and somatostatin levels, as well as arginine-stimulated levels of islet cell hormones).

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age and older.
* Tissue-confirmed diagnosis of pancreatic adenocarcinoma.
* Scheduled for surgical resection of the adenocarcinoma (Whipple or distal pancreatectomy).
* Able to give informed consent

Exclusion Criteria:

* History of any radiation therapy to the abdomen prior to surgery.
* Any contraindication to MRI, including but not limited to implanted metal devices (e.g. pacemaker, berry aneurysm clips, neural stimulator, cochlear implants, or metal in the eye).
* Treatment with an investigational drug within 1 month prior to the day of the study drug administration.
* Current enrollment in any other interventional study.
* Creatinine greater than 2.0.
* Significant liver disease, liver masses, or evidence of portal hypertension.
* Pregnancy.
* History of sensitivity to secretin.
* Unwilling or unable to sign informed consent.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2007-09; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Percent of duct volume change of patients with bicarbonate concentration of duodenal fluid aspirate or acid steatocrit | 12 months
  Our primary aim is to compare S-MRCP with either Endoscopic Pancreatic Function Test (ePFT) (in those patients who undergo esophagogastroduodenoscopy [EGD] or endoscopic ultrasound [EUS]) or acid steatocrit. The primary outcome will be the correlation between duodenal filling on SMRCP (expressed as percent of duct volume change from baseline and maximal values following secretin administration) with either 1) maximal bicarbonate concentration of duodenal fluid aspirate or 2) acid steatocrit (a measure of steatorrhea, expressed as volumetric percentage).

SECONDARY OUTCOMES:
Percentage diameter change on S-MRCP of patients with pancreatic insufficiency | 12 months
  In those patients who are undergoing endocrine pancreatic testing, our secondary aim is to investigate the relationship between other radiological parameters, including percentage diameter change on S-MRCP, with other clinical markers of pancreatic insufficiency, including fecal elastase-1 and vitamin levels, patients' grading of abdominal symptoms, quality-of-life questionnaire scores, and body mass index (BMI).
Pancreatic duct mean diameter of patients with high arginine-stimulated hormone levels | 12 months
  Another secondary aim will be to evaluate MRI imaging parameters (primarily maximal gadolinium signal enhancement, but also non-enhancement measures such as total volume and mean T1 signal) with arginine-stimulated hormone levels (primarily arginine-stimulated insulin levels, but we will also be examining glucagon, amylin, somatostatin and Cpeptide levels).

CONTACTS AND LOCATIONS:
Overall Officials: Harold Frucht, MD, Principal Investigator — Columbia University
Locations (1):
- Columbia University Medical Center, New York, New York, United States